CLINICAL TRIAL: NCT01548118
Title: A Blind, Randomized and Placebo-controlled Clinical Trial With Recombinant HumanPapillomavirus Bivalent (Types 16 and 18) Vaccine (Yeast) in Health Women-Phase I
Brief Title: Evaluate the Safety of Recombinant Human Papillomavirus Bivalent (Types 16 and 18) Vaccine (Yeast) in Healthy Females
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Zerun Biotechnology Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 311-HPV-1001
Record Dates: First submitted 2012-02-29; First posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Human Papillomavirus
Keywords: Human papillomavirus; vaccine; cervical infection; cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Adult Group 1, HPV vaccine 0.5ml (Experimental): 20 women between 18-45 yeas of age, receiving 0,2,6 month-schedule of 0.5ml experimental HPV vaccines.
  Interventions: Biological: HPV 16/18 vaccine, 0,5ml
- Adult Group 1, Placebo 0.5ml (Placebo Comparator): 20 women between 18-45 yeas of age, receiving 0,2,6 month-schedule of 0.5ml aluminum phosphate.
  Interventions: Biological: Placebo control, 0.5ml
- Adult Group 2, HPV vaccine 1.0ml (Experimental): 20 women between 18-45 yeas of age, receiving 0,2,6 month-schedule of 1.0ml experimental HPV vaccines.
  Interventions: Biological: HPV 16/18 vaccine, 1.0ml
- Adult Group 2, Placebo 1.0ml (Placebo Comparator): 20 women between 18-45 yeas of age, receiving 0,2,6 month-schedule of 1.0ml aluminum phosphate.
  Interventions: Biological: Placebo control, 1.0ml
- Children Group 1, HPV vaccine 0.5ml (Experimental): 20 girls between 9-17 yeas of age, receiving 0,2,6 month-schedule of 0.5ml experimental HPV vaccines.
  Interventions: Biological: HPV 16/18 vaccine, 0,5ml
- Children Group 1, Placebo 0.5ml (Placebo Comparator): 20 girls between 9-17 yeas of age, receiving 0,2,6 month-schedule of 0.5ml aluminum phosphate.
  Interventions: Biological: Placebo control, 0.5ml
- Children Group 2, HPV vaccine 1.0ml (Experimental): 20 girls between 9-17 yeas of age, receiving 0,2,6 month-schedule of 1.0ml experimental HPV vaccines.
  Interventions: Biological: HPV 16/18 vaccine, 1.0ml
- Children Group 2, Placebo 1.0ml (Placebo Comparator): 20 girls between 9-17 yeas of age, receiving 0,2,6 month-schedule of 1.0ml aluminum phosphate.
  Interventions: Biological: Placebo control, 1.0ml

INTERVENTIONS:
Biological: HPV 16/18 vaccine, 0,5ml — Subjects were planned to receive HPV vaccine 0.5ml administered intramuscularly according to a 0, 2, 6 month vaccination schedule
  Arms: Adult Group 1, HPV vaccine 0.5ml; Children Group 1, HPV vaccine 0.5ml
Biological: Placebo control, 0.5ml — Subjects were planned to receive three doses of the placebo control 0.5ml administered intramuscularly according to a 0, 2, 6 month vaccination schedule.
  Arms: Adult Group 1, Placebo 0.5ml; Children Group 1, Placebo 0.5ml
Biological: HPV 16/18 vaccine, 1.0ml — Subjects were planned to receive HPV vaccine 1.0ml administered intramuscularly according to a 0, 2, 6 month vaccination schedule
  Arms: Adult Group 2, HPV vaccine 1.0ml; Children Group 2, HPV vaccine 1.0ml
Biological: Placebo control, 1.0ml — Subjects were planned to receive three doses of the placebo control 1.0ml administered intramuscularly according to a 0, 2, 6 month vaccination schedule.
  Arms: Adult Group 2, Placebo 1.0ml; Children Group 2, Placebo 1.0ml

SUMMARY:
This study will evaluate the safety of a novel recombinant human papillomavirus bivalent ( types 16 and 18 ) vaccine ( Yeast ) with different dose in healthy females between 9-45 years of age at enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female between, and including, 9 and 45 years of age at the time of the first vaccination
* Provide legal identification for for the sake of recruitment.
* Be able to understand and sign informed consent prior to enrollment (For subjects below the legal age of consent, informed consent must be signed by parent(s)/legal guardian(s) in addition).
* Subject must be not pregnant at the enrollment and agree to using adequate contraceptive precautions within 7 months.

Exclusion Criteria:

* History of cervical cancer
* History of severe allergic reaction requiring medical intervention (such as oral and throat swelling, difficulty breathing, hypotension or shock)
* History of allergic to vaccine, or to any ingredient of vaccine.
* History of epilepsy, seizures or convulsions, or family history of mental illness
* Subjects are immunocompromised or have been diagnosed as suffering from congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis inflammation (JRA), inflammatory bowel disease or other autoimmune diseases, administration of immunosuppressants with six months prior to the first vaccine dose.
* History of asthma, thyroidectomy, angioneurotic edema, diabetes or malignant
* Asplenia, functional asplenia, or any circumstances result of asplenia or splenectomy
* Medical diagnosis of coagulation abnormalities (eg, clotting factor deficiency, coagulation disorders, platelet anomaly) or obvious bruising or coagulation disorder
* Acute disease or chronic disease acute exacerbation 7 days prior to vaccination
* Administration of immunoglobulins and/or any blood products within 3 months, or administration of any live attenuated vaccine within 28 days, or administration of any subunit or inactivated vaccines within 14 days.
* Fever or axillary temperature> 37.0 °C before vaccination
* During menstrual period, breastfeeding, pregnancy(pregnancy test positive), or planned pregnant within 7 month
* History of hypertension, physical examination systolic blood pressure> 150mmHg and/or diastolic blood pressure> 100mmHg
* Abnormal laboratory tests parameters
* Any clinical significant disease or findings during study screening that, in the opinion of the Investigator may interfere with the study

Ages: 9 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence, intensity and relationship to vaccination of any solicited local or systemic reactions. | 7 days after each vaccine dose
Occurrence, intensity and relationship to vaccination of any unsolicited symptom. | 30 days after finish vaccinations

SECONDARY OUTCOMES:
Neutralizing antibody responses of HPV 16/18 after each vaccine dose. | 30 days after finish vaccinations

CONTACTS AND LOCATIONS:
Overall Officials: Yan-ping Li, MD, Principal Investigator — Guangxi Centers for Disease Control and Prevention
Locations (1):
- GuangXi Center for Diseases Control and Prevention, Nanning, Guangxi, China